CLINICAL TRIAL: NCT05670249
Title: Decompressive Craniectomy In Patients With Malignant Cerebellar Infarction: A Randomized, Controlled Trial in a Turkish Population (DEMCI Trial)
Brief Title: Decompressive Craniectomy in Patients With Cerebellar Infarction
Acronym: DEMCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Emre Kumral, Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EU0691
Record Dates: First submitted 2022-11-20; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Cerebellar Stroke

STUDY DESIGN:
Intervention Model Description: Participants assigned to either conservative medical or SDC group with a 1:1 allocation assignment using a random number table by co-decision of a neurologist, neurosurgeon and statistician
Who Masked: Care Provider
Masking Description: a senior neurologist (E.K. or M.D.) who was not involved in screening, randomization, or patient care, blinded to the therapeutic arm assignment of the patient assessed the mRS (primary outcome), Barthel Index, NIHSS (National Institute of Health Stroke Scale), and SF-36 (secondary outcomes) scores
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical plus medical treatment (Active Comparator): Decompressive surgery protocol was kept constant throughout the study period and defined the following surgical interventions: (1) extensive bilateral suboccipital decompresive craniectomy with duraplasty, optional resection of the posterior arch of atlas, (2) preceding insertion of an external ventricular drainage (EVD) in all cases, and (3) evacuation of necrotic tissue.
  Interventions: Procedure: suboccipital decompressive craniectomy
- conservative medical treatment (No Intervention): Control group (conservative medical) was treated equally aggressive with regard to intensive care measures. Medical management generally followed the Turkish and European guidelines on acute stroke care valid at the time of patient admission.

INTERVENTIONS:
Procedure: suboccipital decompressive craniectomy — extensive bilateral suboccipital decompressive craniectomy with duraplasty
  Other Names: space occupying surgey
  Arms: surgical plus medical treatment

SUMMARY:
The investigators aimed to evaluate the outcome in participants up to 80 years of age with space-occupying cerebellar infarction treated with suboccipital decompressive craniectomy (SDC) compared to medical therapy alone.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, controlled, clinical trial based on a stroke center. The primary end point was survival with favorable outcome, defined as a score of 0 to 3 on the mRS at 12 months (±30 days) after randomization (defined by a score of 0 to 3 on the modified Rankin scale (mRS), which ranges from 0 [no symptoms] to 6 [death]). Secondary outcomes included death, Barthel Index, baseline stroke severity NIHSS (National Institute of Health Stroke Scale), and SF-36 at 6 months and 1-year after randomization. The variables for subgroup analysis were age, sex, time to randomization, lesion volume, brainstem involvement, hemorrhagic transformation.

ELIGIBILITY:
Inclusion Criteria:

* The presence of cerebellar territory infarction with an NIHSS score ≥8.
* Initial Glasgow Coma Scale (GCS) score <9 on admission and clinical deterioration (a score of ≥ 1 decrease on GCS score) within 48 hours from onset.
* Decrease in the level of consciousness to a score of ≥ 1 on item 1a (level of consciousness) of the NIHSS, rapid deterioration to coma.

Exclusion Criteria:

* Prestroke mRS score ≥2.
* Prestroke score on the Barthel Index <95.
* Score on the Glasgow Coma Scale ≤6.
* Both pupils fixed and dilated.
* Any other coincidental brain lesion that might affect outcome.
* Space-occupying hemorrhagic transformation of the infarct.
* Pregnancy.
* Life expectancy <3 years.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The primary end point was survival with favorable outcome, defined as a score of 0 to 3 modified Rankin score | one year
  The modified Rankin scale (mRS), which ranges from 0 [no symptoms] to 6 [death]).

SECONDARY OUTCOMES:
Death | 1 year
  Patient who died due to surgery
Barthel Index, | 1 year
  Barthel index which ranges from 0 [dependent] to 100 [Totally independent)
NIHSS (National Institute of Health Stroke Scale) | 1 year
  independent), NIHSS ranges from 0 to 42 (the higher the score, the more severe the stroke)

IPD SHARING:
Plan to Share IPD: Undecided
Plan to Share IPD is 'Yes"